CLINICAL TRIAL: NCT01769378
Title: A Randomized, Parallel-Arm, Double-Blinded Study Comparing the Effect of Once-Weekly Dulaglutide With Placebo in Patients With Type 2 Diabetes Mellitus on Sulfonylurea Therapy (AWARD-8: Assessment of Weekly AdministRation of LY2189265 in Diabetes - 8)
Brief Title: Study of How Dulaglutide Compares to Placebo in Participants With Type 2 Diabetes Who Are Also on Sulfonylurea Therapy (AWARD-8)
Acronym: AWARD-8
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13193; H9X-MC-GBDG (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Results first posted 2015-10-14 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2015-12

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo administered subcutaneously (SQ) once weekly for 24 weeks added to the participant's prescribed glimepiride dose.
  Interventions: Drug: Placebo; Drug: Glimepiride
- Dulaglutide (Experimental): Dulaglutide 1.5 milligram (mg) administered SQ once weekly for 24 weeks added to the participant's prescribed glimepiride dose.
  Interventions: Drug: Dulaglutide; Drug: Glimepiride

INTERVENTIONS:
Drug: Placebo — Administered SQ
  Arms: Placebo
Drug: Dulaglutide — Administered SQ
  Other Names: LY2189265
  Arms: Dulaglutide
Drug: Glimepiride — Administered PO

SUMMARY:
The purpose of this study is to assess the efficacy and safety of once-weekly dulaglutide compared to placebo in participants with type 2 diabetes who have inadequate glycemic control with sulfonylurea monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Stable dose of sulfonylurea that is at least 50% of the maximum approved dose per the local label for at least 3 months prior to the first study visit
* Have an HbA1c value of ≥7.5% and ≤9.5%, as determined by the central laboratory draw performed at the first study visit
* Accept continued treatment with sulfonylurea therapy, throughout the trial, as required per protocol
* Men and nonpregnant women aged ≥18 years
* Stable weight (±5%) ≥3 months prior to screening
* Body Mass Index (BMI) ≤45 kilograms per square meter (kg/m^2)

Exclusion Criteria:

* Have type 1 diabetes mellitus
* Have been treated with ANY other antihyperglycemic medications (other than sulfonylurea) at the time of the first study visit or within 3 months prior to the first study visit
* Have used insulin therapy (outside of pregnancy) any time in the past 2 years, except for short-term treatment of acute conditions, and up to a maximum of 4 weeks; any insulin within 3 months prior to the first study visit is exclusionary
* Have been treated with drugs that promote weight loss within 3 months prior to the first study visit
* Are receiving chronic (>14 days) systemic glucocorticoid therapy or have received such therapy within the 4 weeks immediately prior to the first study visit
* Have had any of the following Cardiovascular (CV) conditions within 2 months prior to the first study visit: acute myocardial infarction, New York Heart Association Class III or Class IV heart failure, or cerebrovascular accident
* Have a known clinically significant gastric emptying abnormality (eg, severe diabetic gastroparesis or gastric outlet obstruction) or have undergone gastric bypass (bariatric) surgery or restrictive bariatric surgery
* Have acute or chronic hepatitis, signs and symptoms of any other liver disease, or alanine transaminase level >2.5 times the upper limit of normal
* Have a history of chronic pancreatitis or acute idiopathic pancreatitis, or were diagnosed with any type of acute pancreatitis within the 3 month period prior to the first study visit
* Have an estimated glomerular filtration rate [eGFR] <30 milliliter per minute per 1.73 square meter (mL/min/1.73 m^2), calculated using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation as determined by the central laboratory at the first study visit
* Have any self or family history of type 2A or type 2B multiple endocrine neoplasia (MEN 2A or 2B) in the absence of known C-cell hyperplasia (this exclusion includes those participants with a family history of MEN 2A or 2B, whose family history for the syndrome is Rearranged during Transfection (RET) negative; the only exception for this exclusion will be for participants whose family members with MEN 2A or 2B have a known RET mutation and the potential participant for the study is negative for that RET mutation)
* Have any self or family history of medullary C-cell hyperplasia, focal hyperplasia, carcinoma (including sporadic, familial or part of MEN 2A or 2B syndrome)
* Have a serum calcitonin ≥20 picogram per milliliter (pg/mL) as determined by the central laboratory at the first study visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (31):
- United States (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chino, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trenton, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Bronx, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beaver, Pennsylvania
- Argentina (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Corrientes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosario
- Austria (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salzburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zams
- Croatia (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krapinske Toplice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osijek
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rijeka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Slavonski Brod
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Varaždin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zagreb
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampico
- Romania (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alba Iulia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Galati
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oradea
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sibiu
- Slovenia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Celje
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ljubljana
- South Africa (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloemfontein
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durban
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Somerset West

REFERENCES:
- [Derived] Ferdinand KC, Dunn J, Nicolay C, Sam F, Blue EK, Wang H. Weight-dependent and weight-independent effects of dulaglutide on blood pressure in patients with type 2 diabetes. Cardiovasc Diabetol. 2023 Mar 9;22(1):49. doi: 10.1186/s12933-023-01775-x. PMID 36894938

RESULTS

PARTICIPANT FLOW:
Groups:
- Dulaglutide: Dulaglutide 1.5 milligram (mg) administered subcutaneously (SQ) once weekly for 24 weeks added to the participant's prescribed glimepiride dose.
- Placebo: Placebo administered SQ once weekly for 24 weeks added to the participant's prescribed glimepiride dose.
Period: Overall Study
Arm/Group | Dulaglutide | Placebo
Started | 240 | 60
Received at Least 1 Dose of Study Drug | 239 | 60
Completed | 215 (Completed the study on study treatment) | 56 (Completed the study on study treatment)
Not Completed | 25 | 4
Not completed — Adverse Event | 10 | 0
Not completed — Entry criteria not met | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 10 | 3
Not completed — Sponsor Decision | 1 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population: all randomized participants who received at least one dose of study drug.
Groups:
- Dulaglutide: Dulaglutide 1.5 mg administered SQ once weekly for 24 weeks added to the participant's prescribed glimepiride dose.
- Total: Total of all reporting groups
Arm/Group | Dulaglutide | Placebo | Total
Number analyzed (Participants) | 239 | 60 | 299
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 182 | 49 | 231
  >=65 years | 57 | 11 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.73 (10.20) | 58.23 (7.40) | 57.83 (9.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 32 | 167
  Male | 104 | 28 | 132
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 112 | 27 | 139
  Not Hispanic or Latino | 127 | 33 | 160
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 21 | 5 | 26
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 4 | 11
  White | 202 | 47 | 249
  More than one race | 6 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 29 | 8 | 37
  Austria | 4 | 1 | 5
  Romania | 78 | 18 | 96
  United States | 57 | 14 | 71
  South Africa | 7 | 3 | 10
  Mexico | 40 | 10 | 50
  Slovenia | 13 | 3 | 16
  Croatia | 9 | 2 | 11
  Puerto Rico | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin A1c (HbA1c) at 24 Weeks
Description: Least Squares Means (LS Means) of the HbA1c change from baseline to primary endpoint was adjusted by fixed effects of treatment, country, visit, treatment-by-visit interaction, participant as random effect and baseline HbA1c as covariate, via a Mixed-effects model for repeated measures (MMRM) analysis using restricted maximum likelihood (REML).
Time Frame: Baseline, 24 Weeks
Population: Participants who were randomized and received at least one dose of study drug with evaluable HbA1c data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: percent change of HbA1c
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 215 | 53
percent change of HbA1c | -1.38 (0.08) | -0.11 (0.14)
Statistical Analysis 1: Comparison: Dulaglutide vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Squares Mean Difference = -1.27, 95% CI 2-sided [-1.57 to -0.97], Standard Error of Mean 0.15

2. Secondary Outcome: Percentage of Participants Who Achieve HbA1c <7.0% and ≤6.5% at 24 Weeks
Description: The percentage of participants who achieved the target HbA1c values at endpoint will be analyzed with a repeated logistic regression model (the generalized estimation equation [GEE] model). The model includes country, treatment, visit and treatment interaction and baseline HbA1c as a continuous covariate.
Time Frame: 24 Weeks
Population: Participants who were randomized and received at least one dose of study drug with evaluable HbA1c data.
Measure: Number; unit: percentage of participants
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 215 | 53
percentage of participants
  Percent Achieved <7.0 HbA1c Level | 55.3 | 18.9
  Percent Achieved ≤6.5 HbA1c Level | 40.0 | 9.4
Statistical Analysis 1: Comparison: Dulaglutide vs Placebo; <7.0% HbA1c; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Sequential gatekeeping strategy was used to adjust for multiplicity; Odds Ratio (OR) = 11.37, 95% CI 2-sided [3.82 to 33.84]
Statistical Analysis 2: Comparison: Dulaglutide vs Placebo; ≤6.5% HbA1c; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 11.45, 95% CI 2-sided [3.71 to 35.34]

3. Secondary Outcome: Change From Baseline in Fasting Serum Glucose (FSG) at 24 Weeks
Description: LS Means of the FSG from baseline to primary endpoint was adjusted by fixed effects of treatment, country, baseline HbA1c strata, and baseline FSG as covariate, via Analysis of Covariance Model (ANCOVA) with Last Observation Carried Forward (LOCF).
Time Frame: Baseline, 24 Weeks
Population: Participants who received at least one dose of study drug and had evaluable FSG data at both baseline and post-baseline. LOCF was used to impute missing post-baseline values. If no data after date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 218 | 51
milligrams per deciliter (mg/dL) | -30.60 (4.46) | 2.93 (6.76)
Statistical Analysis 1: Comparison: Dulaglutide vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Sequential gatekeeping strategy was used to adjust for multiplicity; Least Squares Mean Difference = -33.54, 95% CI 2-sided [-46.55 to -20.53], Standard Error of Mean 6.60

4. Secondary Outcome: Change From Baseline in Body Weight at 24 Weeks
Description: LS Means of the body weight change from baseline to primary endpoint was adjusted by fixed effects of treatment, country, visit, treatment-by-visit interaction, participant as random effect and baseline body weight as covariate, via a MMRM analysis using REML.
Time Frame: Baseline, 24 Weeks
Population: Participants who received at least one dose of study drug and had evaluable body weight data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 212 | 53
kilograms (kg) | -0.91 (0.21) | -0.24 (0.40)
Statistical Analysis 1: Comparison: Dulaglutide vs Placebo; Test type: Superiority or Other; p = 0.120, Mixed Models Analysis; Sequential gatekeeping strategy was used to adjust for multiplicity; Least Squares Mean Difference = -0.68, 95% CI 2-sided [-1.53 to 0.18], Standard Error of Mean 0.43

5. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at 24 Weeks
Description: LS Means of the BMI change from baseline to primary endpoint was adjusted by fixed effects of treatment, country, visit, treatment-by-visit interaction, participant as random effect and baseline BMI as covariate, via a MMRM analysis using REML.
Time Frame: Baseline, 24 Weeks
Population: Participants who received at least one dose of study drug and evaluable BMI data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: kilograms per/square meter kg/m^2
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 212 | 53
kilograms per/square meter kg/m^2 | -0.32 (0.08) | -0.10 (0.15)
Statistical Analysis 1: Comparison: Dulaglutide vs Placebo; Test type: Superiority or Other; p = 0.161, Mixed Models Analysis — No adjustment for multiplicity; Least Squares Mean Difference = -0.23, 95% CI 2-sided [-0.54 to 0.09], Standard Error of Mean 0.16

6. Secondary Outcome: Change From Baseline in Mean of All 7-Point Self Monitored Plasma Glucose (SMPG) at 24 Weeks
Description: LS Means of the SMPG change from baseline to primary endpoint at week 24 was adjusted by fixed effects of treatment, country, visit, treatment-by-visit interaction, participant as random effect and baseline SMPG value as covariate, via a MMRM analysis using REML.
Time Frame: Baseline, 24 Weeks
Population: Participants who received at least one dose of study drug and had evaluable SMPG data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 203 | 49
mg/dL | -37.22 (3.10) | -8.27 (4.77)
Statistical Analysis 1: Comparison: Dulaglutide vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -28.95, 95% CI 2-sided [-38.49 to -19.40], Standard Error of Mean 4.85

7. Secondary Outcome: Number of Participants With Reported and Adjudicated Cardiovascular Events
Description: Information on cardiovascular (CV) risk factors was collected at baseline. Deaths and nonfatal cardiovascular adverse events (AEs) were adjudicated by an external committee of physicians with cardiology expertise. Nonfatal cardiovascular AEs to be adjudicated included myocardial infarction, hospitalization for unstable angina, hospitalization for heart failure, coronary interventions, and cerebrovascular events, including cerebrovascular accident (stroke) and transient ischemic attack. The number of participants with CV events confirmed by adjudication is summarized cumulatively at 24 weeks plus 30-day follow up. Serious and all other non-serious adverse events regardless of causality are summarized in the Reported Adverse Events module.
Time Frame: Baseline through 24 Weeks, 30-day Follow Up
Population: ITT population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 239 | 60
participants
  Any reported CV events | 2 | 0
  Any adjudicated nonfatal CV events | 2 | 0
  Any confirmed adjudicated CV deaths | 0 | 0

8. Secondary Outcome: Number of Participants With Adjudicated Acute Pancreatitis Events
Description: The number of participants with pancreatitis confirmed by adjudication is summarized cumulatively at 24 weeks plus 30-day follow up. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 24 Weeks, 30-day Follow Up
Population: ITT population: all randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 239 | 60
participants | 0 | 0

9. Secondary Outcome: Change From Baseline in Calcitonin at 24 Weeks
Time Frame: Baseline, 24 Weeks
Population: Participants who received at least one dose of study drug and evaluable calcitonin data at baseline and post-baseline.
Measure: Median (Inter-Quartile Range); unit: picogram per milliliter (pg/ml)
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 215 | 59
picogram per milliliter (pg/ml) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

10. Secondary Outcome: Percentage of Participants With Self-Reported Events of Hypoglycemia
Description: Hypoglycemic events (HE) were classified as severe (defined as episodes requiring the assistance of another person to actively administer resuscitative actions), documented symptomatic (defined as any time a participant feels that he/she is experiencing symptoms and/or signs associated with hypoglycemia, and has a plasma glucose level of =<3.9 mmol/L), asymptomatic (defined as events not accompanied by typical symptoms of hypoglycemia but with a measured plasma glucose of =<3.9 mmol/L), nocturnal (defined as any hypoglycemic event that occurred between bedtime and waking), or probable symptomatic (defined as events during which symptoms of hypoglycemia were not accompanied by a plasma glucose determination). Percentage is calculated as the number of participants reporting HE each visit/ the total number of participants reporting HE during the entire study treatment period.
Time Frame: Baseline through 24 Weeks
Population: ITT Population: all randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 239 | 60
percentage of participants
  Symptomatic | 11.3 | 1.7
  Asymptomatic | 13.4 | 1.7
  Probable | 2.5 | 0.0
  Severe | 0 | 0
  Nocturnal | 6.7 | 1.7

11. Secondary Outcome: Rate of HE Adjusted Per 30 Days
Description: The hypoglycemia rate per 30 days during defined period is calculated by the number of hypoglycemia events within the period/number of days participant at risk within the period*30 days.
Time Frame: Baseline through 24 weeks
Population: ITT population: all randomized participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: number of events/participants/30 days
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 239 | 60
number of events/participants/30 days
  Total HE | 0.19 (0.59) | 0.01 (0.03)
  Documented symptomatic HE | 0.07 (0.33) | 0.00 (0.02)
  Asymptomatic HE | 0.11 (0.45) | 0.00 (0.02)
  Severe HE | 0 (0.0) | 0 (0.0)
  Nocturnal HE | 0.02 (0.16) | 0.00 (0.02)
  Probable symptomatic HE | 0.01 (0.04) | 0 (0.0)

12. Secondary Outcome: Percentage of Participants Requiring Additional Intervention for Severe, Persistent Hyperglycemia
Description: Additional Intervention: any additional therapeutic intervention in participants who developed persistent, severe hyperglycemia despite full compliance with the assigned therapeutic regimen, or initiation of an alternative antihyperglycemic medication following study drug discontinuation.
Time Frame: Baseline through 24 Weeks
Population: ITT population: all randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 239 | 60
percentage of participants | 2.1 | 11.7

13. Secondary Outcome: Time to Initiation of Additional Intervention for Severe, Persistent Hyperglycemia
Description: An additional intervention (rescue therapy) was defined as any additional therapeutic intervention in participants who developed persistent, severe hyperglycemia despite full compliance with the assigned therapeutic regimen, or initiation of an alternative antihyperglycemic medication following study drug discontinuation. Participants who had no rescue therapy within specified study period were considered as censored observations at the last available contact date up to specified study period.
Time Frame: Baseline through 24 Weeks
Population: ITT population: All randomized participants who received at least one dose of study drug.
Measure: Mean (Standard Error); unit: weeks
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 239 | 60
weeks | 22.59 (0.36) | 22.47 (0.66)

14. Secondary Outcome: Dulaglutide Anti-Drug Antibodies (ADA)
Description: Number of participants with treatment emergent (TE) dulaglutide anti-drug antibodies from postbaseline to follow up were summarized. A participant is considered to have TE dulaglutide ADA if the participant has at least one titer that is treatment-emergent relative to baseline, defined as a 4-fold or greater increase in titer from baseline measurement.
Time Frame: Baseline up to 4 Weeks Post-Last Dose of Study Drug
Population: ITT population: all randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Dulaglutide
Number analyzed (Participants) | 239
participants | 2

15. Secondary Outcome: Change From Baseline in Lipase
Description: A summary of changes in lipase evaluation from baseline to endpoint.
Time Frame: Baseline, 24 Weeks
Population: All participants who received at least one dose of study drug and had evaluable lipase data at both baseline and post-baseline. LOCF was used to impute missing postbaseline values. If no data after date of randomization, the endpoint was considered missing.
Measure: Median (Inter-Quartile Range); unit: Units/Liter
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 233 | 60
Units/Liter | 8.0 [1.0 to 18.0] | 4.5 [-2.5 to 15.5]

16. Secondary Outcome: Change From Baseline in Amylase
Description: A summary of changes in amylase evaluation from baseline to endpoint.
Time Frame: Baseline, 24 Weeks
Population: Participants who received at least one dose of study drug and had evaluable amylase data at both baseline and post-baseline. LOCF was used to impute missing postbaseline values. If no data after date of randomization, the endpoint was considered missing.
Measure: Median (Inter-Quartile Range); unit: Units/Liter
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 233 | 60
Units/Liter | 8.0 [1.0 to 18.0] | 2.0 [-5.0 to 11.0]

ADVERSE EVENTS:
Arm/Group | Dulaglutide | Placebo
Serious Adverse Events (participants affected / at risk) | 9/239 | 0/60
Other Adverse Events (participants affected / at risk) | 44/239 | 3/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dulaglutide (N=239) | Placebo (N=60)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dulaglutide (N=239) | Placebo (N=60)
Diarrhoea (Gastrointestinal disorders) | 20 (30) | 0 (0)
Eructation (Gastrointestinal disorders) | 14 (24) | 0 (0)
Nausea (Gastrointestinal disorders) | 25 (31) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days